CLINICAL TRIAL: NCT01580384
Title: A Non-Drug Study of The Suitability of Neurocognitive Tests And Functioning Scales For The Measurement of Cognitive And Functioning Changes in Individuals With Down Syndrome
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: BP25612
Record Dates: First submitted 2012-03-23; First posted 2012-04-19 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-03

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This non-drug, longitudinal, multi-center, multi-national study will evaluate the suitability of neurocognitive tests and functioning scales for the measurement of cognitive and functioning changes in individuals with Down Syndrome. Tests will be administered at clinic visits in Weeks 1, (4) and 24. The duration of the study for each individual will be between 24 and 27 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 12 to 30 years of age, with diagnosis of Down Syndrome
* Down Syndrome subjects meeting clinical diagnostic criteria for generalized anxiety disorders, major depressive disorders, autism spectrum disorder, attention deficit and hyperactivity disorder can participate in the study provided they are on stable medication for at least 8 weeks prior to screening and likely to cooperate and take part successfully in the study assessments

Exclusion Criteria:

* Subjects with DSM-IV axis I and II psychiatric disorders, except those authorized in the inclusion criteria
* Subjects who may not be able to comply with the protocol or perform the outcome measures due to significant hearing or visual impairment
* Subjects with evidence of dementia or meeting clinical diagnosis for dementia
* Subjects with thyroid dysfunction or diabetes that is not adequately controlled and stabilized on treatment for at least 8 weeks prior to randomization

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Individuals with Down Syndrome
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2012-02; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Neurocognitive batteries/tests/scales: Suitability for individuals with Down syndrome assessed by number of tests completed/subjects completing, ceiling/floor effect, variance estimate of baseline/change from baseline | approximately 1.5 years

SECONDARY OUTCOMES:
Test/re-test reliability: Changes in test results over 4 weeks | approximately 1.5 years
Changes in test results over 6 month interval | approximately 1.5 years
Correlations between test results on functioning, adaptive behavior and cognition and IQ level | approximately 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (12):
- United States (2):
  - Tucson, Arizona
  - Durham, North Carolina
- Argentina (2):
  - Ciudad Autonoma de Bs As
  - Ciudad de Buenos Aires
- Kentville, Nova Scotia, Canada
- France (2):
  - Paris
  - Saint-Etienne
- Italy (2):
  - Rome, Lazio
  - Palermo, Sicily
- Barcelona, Barcelona, Spain
- United Kingdom (2):
  - London
  - Redruth

REFERENCES:
- [Derived] Spiridigliozzi GA, Goeldner C, Edgin J, Hart SJ, Noeldeke J, Squassante L, Visootsak J, Heller JH, Khwaja O, Kishnani PS, Liogier d'Ardhuy X. Adaptive behavior in adolescents and adults with Down syndrome: Results from a 6-month longitudinal study. Am J Med Genet A. 2019 Jan;179(1):85-93. doi: 10.1002/ajmg.a.60685. Epub 2018 Dec 20. PMID 30569586